CLINICAL TRIAL: NCT05969561
Title: Ultrasound-Guided Femoral Nerve Block
Brief Title: Emergency Physician-performed Ultrasound-guided Femoral Nerve Blocks in Patients With Hip Fractures.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 202211021RINB
Record Dates: First submitted 2023-07-23; First posted 2023-08-01 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-06

CONDITIONS: Hip Fractures
Keywords: Ultrasound-guided femoral nerve block
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ultrasound-guided femoral nerve block (Active Comparator): Patients with hip fractures had underwent Ultrasound-guided femoral nerve block performed by emergency physicians.
  Interventions: Procedure: ultrasound-guided femoral nerve block
- The liberal use of pain medication (Sham Comparator): Patients with hip fractures had given intravenous or intramuscular opioids or NSAID at the emergency department.
  Interventions: Drug: Intravenous or intramuscular pain medication

INTERVENTIONS:
Procedure: ultrasound-guided femoral nerve block — The local analgesia is injected and infiltrated around the femoral nerve under ultrasound guidance.
  Arms: Ultrasound-guided femoral nerve block
Drug: Intravenous or intramuscular pain medication — Intravenous or intramuscular pain medication is given for patients with hip fracture.
  Arms: The liberal use of pain medication

SUMMARY:
In this prospective study, emergency physicians perform ultrasound-guided femoral nerve block for patients with hip fractures. We compare the effectiveness of analgesia and patient satisfaction of ultrasound-guided femoral nerve block with liberal use of the pain medicine in the emergency department. The primary outcome is the assessment of time to relief the pain with fewer adverse effects and less rescue pain medication use. The secondary outcome is patient satisfaction and adverse effects for different method of pain control.

DETAILED DESCRIPTION:
The aim of this study is to compare the effectiveness of ultrasound-guided femoral nerve blocks performed by emergency physicians for pain control in the emergency department with traditional pain medicine.

This study is a prospective before-and-after design. The enrollees are 20-year-old and older adult patients with hip fractures. We use numerical rating scale using a 0-10 scale to assess pain severity at the different time frame after giving pain medicine. The scale zero means "no pain" and scale 10 means "the worst pain imaginable".

The primary outcome is assessed by the reduction of pain scale which are taken on a numeric rating scale every 30 minutes before and after pain management. The secondary outcome compares complications, adverse effects and patient satisfaction for different method of pain control.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 20-year-old with hip fractures
* Stay in the emergency department for at lease two hours

Exclusion Criteria:

* hemodynamic unstable
* major trauma in addition to hip fractures
* the use of any pain management before the arrival of emergency department
* chronic opioid use
* inability to understood the numerical rating scale after instruction
* allergy to local anesthetics
* coagulopathy
* injection site infection

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-07-03 (Actual); Primary Completion 2025-03-05 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
a short time of pain relief | 2 hours
  The numerical pain score from 0 to 10 is used to assess pain severity and the scale 0 means no pain and the scale 10 means the worst pain imaginable. The pain score assessed for the leg with hip fracture at rest and with movement will be recorded after different pain medicine and the reduction of pain score at different time frame will be evaluated. The more reduction of pain score, the better.

SECONDARY OUTCOMES:
Adverse effects | two hours
  Any adverse effects of different pain medication
Patient satisfaction | two hours
  The difference of patient satisfaction between ultrasound-guided femoral nerve block and the liberal use of pain medication
Complications of ultrasound-guided femoral nerve block | two hours and one week after ultrasound-guided femoral nerve block or after hospital discharge
  Any complications of ultrasound-guided femoral nerve block

CONTACTS AND LOCATIONS:
Locations (1):
- NTUH Yunlin Branch, Douliu, Yunlin County, Taiwan